CLINICAL TRIAL: NCT03221218
Title: Enhanced Screening for Early Treatment Targets After Mild Traumatic Brain Injury
Brief Title: Enhanced Screening for Early Treatment Targets After MTBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Vancouver Coastal Health (Other Government); Fraser Health (Other)
Responsible Party: Principal Investigator, Noah Silverberg, Clinical Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: H17-00584
Record Dates: First submitted 2017-07-12; First posted 2017-07-18 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Brain Concussion
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Patients will be blinded to their group assignment. Family physicians will not be aware that they are involved in a research study until the completion of the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced screening-informed letter (Experimental): Family physicians will receive a letter that includes their patient's screening test results and associated symptom-specific recommendations from the Ontario Neurotrauma Foundation clinical practice guidelines for MTBI (2013).
  Interventions: Other: Enhanced screening-informed follow up letter
- Standard letter (No Intervention): Family physicians will receive a letter that includes generic recommendations for managing MTBI based on the Ontario Neurotrauma Foundation clinical practice guidelines (2013). Screening test results will not be provided.

INTERVENTIONS:
Other: Enhanced screening-informed follow up letter — Family Physicians will be sent a letter that includes their screening test results and associated symptom-specific recommendations from the Ontario Neurotrauma Foundation clinical practice guidelines.
  Arms: Enhanced screening-informed letter

SUMMARY:
The study will examine whether enhancing screening-informed follow-up letters will improve (i) family physician compliance with best practice guidelines for managing persistent symptoms following concussion, and (ii) clinical outcomes from concussion.

DETAILED DESCRIPTION:
Family physicians are well positioned to proactively manage symptoms in the weeks following MTBI, which could prevent chronicity and reduce the need for specialist treatment. Clinical practice guidelines are now available for MTBI management in primary care, such as those developed by the Ontario Neurotrauma Foundation (ONF). However, awareness and use of these guidelines may be low. Distilling the guidelines into a small number of actionable messages that are tailored to an individual patient may facilitate family physician implementation.

The ONF guidelines for MTBI propose that early intervention should prioritize the most readily treatable symptoms - mood (depression and anxiety), insomnia, and headaches. The present cluster randomized trial will evaluate whether screening for these conditions and sending family physicians treatment algorithms for positive screening test results will result in earlier evidence-based treatment.

Patients will be recruited from two concussion clinics that provide group education sessions. Following the education session, eligible participants will complete self-reported screening measures for depression, anxiety, insomnia, and headaches. Family physicians will be randomized to receive these screening test results with associated treatment algorithms from the ONF guidelines or a letter providing generic MTBI management recommendations from the ONF guidelines (currently done as usual care).

Patients will be assessed by telephone one month and three months after the intervention. The primary outcome will be patient-reported treatment utilization that is congruent with the ONF guidelines for depression, anxiety, insomnia, and headaches after MTBI.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 60 years.
* Has a family physician.
* Physician diagnosed MTBI less than 3 months ago.
* English reading comprehension sufficient for the consent form and standardized questionnaires.

Exclusion Criteria:

* English reading comprehension not sufficient for the consent form and standardized questionnaires.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2017-08-09 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2021-06-22 (Actual)

PRIMARY OUTCOMES:
Family physician compliance with guidelines | 1 month after intervention.
  Patient recall of receiving advice, referrals, and prescriptions from their family physician.

SECONDARY OUTCOMES:
Family physician compliance with guidelines (chart review) | 6 to 12 months post injury
  Advice, referrals, and prescriptions related to MTBI care, extracted from chart audits.
Rivermead Post-Concussion Symptoms Questionnaire | 1- and 3-months after intervention.
Generalized Anxiety Disorder-7 (GAD-7) | 1- and 3-months after intervention.
Personal Health Questionnaire-9 (PHQ-9) | 1- and 3-months after intervention.
Insomnia Severity Scale (ISI) | 1- and 3-months after intervention.
World Health Organization Disability Schedule (WHODAS-II) 12 item | 1- and 3-months after intervention.
Quality of Life after Brain Injury Overall Scale (QOLIBRI-OS) | 1- and 3-months after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Noah Silverberg, PhD, Principal Investigator — University of British Columbia
Locations (1):
- GF Strong Rehab Centre, 4255 Laurel Street, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Cassetta BD, Cairncross M, Brasher PMA, Panenka WJ, Silverberg ND. Avoidance and endurance coping after mild traumatic brain injury are associated with disability outcomes. Rehabil Psychol. 2021 May;66(2):160-169. doi: 10.1037/rep0000372. Epub 2020 Dec 31. PMID 33382332
- [Derived] Silverberg ND, Panenka WJ, Lizotte PP, Bayley MT, Dance D, Li LC. Promoting early treatment for mild traumatic brain injury in primary care with a guideline implementation tool: a pilot cluster randomised trial. BMJ Open. 2020 Oct 20;10(10):e035527. doi: 10.1136/bmjopen-2019-035527. PMID 33082178